CLINICAL TRIAL: NCT05497583
Title: Clinical Performance of Acetone Based HEMA-Free Universal Adhesive Versus Isopropanol Based HEMA-Free Universal Adhesive For Restoring Non-Carious Cervical Lesions Over A Period Of 18-Months Follow Up Using FDI Criteria: A Randomized Controlled Trial
Brief Title: HEMA-free Universal Adhesives for Restoring Non-carious Cervical Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hanan Shawky Ramadan, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: universal adhesive
Record Dates: First submitted 2022-08-06; First posted 2022-08-11 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Universal Adhesive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetone based HEMA free Universal Adhesive (Experimental): Patients with non-carious cervical lesions will be treated with Acetone Based HEMA-free Universal Adhesive (BeautiBond universal adhesive ) applied in a self-etch approach with (SE) selective enamel etching.
  Interventions: Other: Acetone based HEMA -free universal Adhesive
- Isopropanol based HEMA-free universal Adhesive (Active Comparator): Patients with non-carious cervical lesions will be treated with isopropanol-based HEMA-free universal Adhesive (Prime&Bond universal™ Adhesive system) applied in a self-etch approach with (SE) selective enamel etching.
  Interventions: Other: Isopropanol based HEMA- free universal Adhesive

INTERVENTIONS:
Other: Acetone based HEMA -free universal Adhesive — Teeth that meet the inclusion criteria will be selected. the operator will prepare incisal bevel. Rubber dam isolation will be used .apply etchant (phosphoric acid etching gel 37 %) only on enamel for 15 s Rinse, for 10 s Air dry to remove excess water then will apply Universal adhesive to the entire bonding surface according to manufacture instructions. Bioactive composite ( beautifill II ) will be used.
  Arms: Acetone based HEMA free Universal Adhesive
Other: Isopropanol based HEMA- free universal Adhesive — Teeth that meet the inclusion criteria will be selected. the operator will prepare incisal bevel. Rubber dam isolation will be used .apply etchant (phosphoric acid etching gel 37 %) only on enamel for 15 s Rinse, for 10 s Air dry to remove excess water then will apply Universal adhesive to the entire bonding surface according to manufacture instructions. resin composite (Neo Spectra™ ST) will be used.
  Arms: Isopropanol based HEMA-free universal Adhesive

SUMMARY:
because of the recent introduction of universal adhesives, little information is currently available about the bond durability of universal adhesives to various substrates. Evaluation of bond durability is important since the stability of the bond between the adhesive and substrates is related to the clinical success of restorations. Because significant hydrolysis of the dentin-resin interface occurs after 6-12 months, a clinical trial of at least 18 months' duration is indicated to more accurately depict the likelihood of long-term clinical success

DETAILED DESCRIPTION:
Cervical restorations are ever challenging because of difficulties in moisture control, caries access, and proximity to the gingival margin. Both mechanical and non-mechanical factors act to hinder the longevity of cervical restoration newer materials are readily introduced in the market with improved chemomechanical properties, longevity, patient safety, and comfort.

The introduction of new-generation adhesive systems has aimed at reducing technique sensitivity and the number of clinical steps required for adhesion. There has been a trend toward the use of less time-consuming options, continuing this trend, universal adhesives have recently been introduced to the profession. However, because of the recent introduction of universal adhesives, little information is currently available about the bond durability of universal adhesives to various substrates. Evaluation of bond durability is important since the stability of the bond between the adhesive and substrates is related to the clinical success of restorations. Although the most reliable conclusions about the performance of adhesives in the oral environment are derived from clinical trials.

To evaluate the effectiveness and clinical performance of adhesive systems, the American Dental Association (ADA) recommends clinical trials on non-carious cervical lesions (NCCLs), as composite resin restorations only remain bonded to these lesions by the micromechanical interlocking produced by the adhesive systems. The immediate, short-term, and long-term bonding performance of adhesive systems are then evaluated by retention, marginal integrity, and marginal discoloration. There are many attempts to improve bonding to substrates, bond strength, and bond durability, one of these attempts is the newly introduced universal adhesive (BeautiBond ).

ELIGIBILITY:
Inclusion Criteria:

* Participants had to be in good general health, be at least 18 years old
* have an acceptable oral hygiene level
* Participants were required to have NCCLs in different teeth preferably anterior or posterior that needed to be restored.
* These lesions had to be noncarious
* deeper than 1 mm
* involve both the enamel and dentin of vital teeth without mobility.

Exclusion Criteria:

* Uncooperative behavior, limits the use of adhesive due to hampering of adequate field or isolation techniques throughout the procedure.
* Patients allergic to the adhesive material. Patients with extremely poor oral hygiene
* severe or chronic periodontitis
* heavy bruxism habits
* Pulp involvement

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Primary outcome (marginal staining) | 18 months
  FDI (World Dental Federation)criteria

SECONDARY OUTCOMES:
Retention, marginal adaptation, Postoperative (Hyper-Sensitivity), and Recurrence of Caries | T0=Baseline immediate postoperative T1= 6 months follow up. T2=12 months follow up. T3=18 months follow up.
  FDI (World Dental Federation)criteria